CLINICAL TRIAL: NCT05819099
Title: The Role of Artificial Intelligence in Endoscopic Diagnosis of Esophagogastric Junctional Adenocarcinoma：A Single Center, Case-control, Diagnostic Study
Status: Not yet recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Other Study IDs: 2023SDU-QILU-1
Record Dates: First submitted 2023-04-06; First posted 2023-04-19 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-04

CONDITIONS: Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training Set
  Interventions: Diagnostic Test: An Intelligent Endoscopic Diagnosis System Developed and Verified Based on Deep Learning
- Test Set
  Interventions: Diagnostic Test: An Intelligent Endoscopic Diagnosis System Developed and Verified Based on Deep Learning
- Verification Set
  Interventions: Diagnostic Test: An Intelligent Endoscopic Diagnosis System Developed and Verified Based on Deep Learning

INTERVENTIONS:
Diagnostic Test: An Intelligent Endoscopic Diagnosis System Developed and Verified Based on Deep Learning — This study will compare the established AI model with the diagnostic results of endoscopists to evaluate the clinical auxiliary value of the model for endoscopists.

SUMMARY:
This is a single center, case-control, diagnostic study.The aim of this study is to use deep learning methods to retrospectively analyze the imaging data of gastrointestinal endoscopy in Qilu Hospital, and construct an artificial intelligence model based on endoscopic images for detecting and determining the depth of invasion of esophagogastric junctional adenocarcinoma.This study will also compare the established AI model with the diagnostic results of endoscopists to evaluate the clinical auxiliary value of the model for endoscopists.The research includes stages such as data collection and preprocessing, artificial intelligence model development, model testing and evaluation. The gastroscopy image dataset constructed by this research institute mainly includes three modes of endoscopic imaging: white light endoscopy, optical enhancement endoscopy (OE), and narrowband imaging endoscopy (NBI).

ELIGIBILITY:
Inclusion Criteria:

* This study included endoscopic images of patients aged 18 and above who underwent endoscopic examination or treatment
* All patients in the case group need to be pathologically confirmed as esophageal gastric junction adenocarcinoma, and a pathologist has conducted a standardized pathological evaluation of the tumor classification of the lesion, including the overall appearance, size, differentiation type, depth of infiltration, presence or absence of lymphatic/vascular invasion, surgical margin status, etc.
* The endoscopic images of the control group patients need to be confirmed by biopsy pathology or at least two experienced endoscopists (with operating experience>5000 cases) to jointly confirm that they have clear benign manifestations

Exclusion Criteria:

* The patient has a previous history of endoscopic treatment or surgery for the esophageal gastric junction.
* Necessary clinical information cannot be provided during the research process (patient age, gender, lesion characteristics, endoscopic manifestations, endoscopic images, etc.)
* Low quality endoscopic images, such as those severely affected by bleeding, aperture, blurring, defocusing, artifacts, or excessive mucus after biopsy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study included endoscopic images of the esophageal gastric junction retrieved from the Endoscopy Center of Qilu Hospital for training and testing the model.The study population underwent pathological examination and the pathological results were used as the gold standard.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2025-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 36 months
  The researchers calculated the sensitivity of the established AI model and compared it with endoscopists of different levels.
Specificity | 36 months
  The researchers calculated the specificity of the established AI model and compared it with endoscopists of different levels.
Negative predictive value | 36 months
  The researchers calculated the negative predictive value of the established AI model and compared it with endoscopists of different levels.
Positive predictive value | 36 months
  The researchers calculated the positive predictive value of the established AI model and compared it with endoscopists of different levels.
Accuracy | 36 months
  The researchers calculated accuracy positive predictive value of the established AI model and compared it with endoscopists of different levels.